CLINICAL TRIAL: NCT06931704
Title: A Multi-center, Open-label, Phase 2 Randomized Study of Elranatamab Plus Lenalidomide Versus Daratumumab Plus Lenalidomide as Post Transplantation Maintenance Therapy in Patients With Newly-diagnosed Myeloma. IFM 2024-06
Brief Title: Comparison of Elranatamab and Lenalidomide Versus Daratumumab and Lenalidomide as Post-transplant Maintenance Therapy in Patients With Newly Diagnosed Myeloma (ElMMA)
Acronym: IFM 2024_06
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC23_0603
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; maintenance; elranatamab; lenalidomide; daratumumab
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care : Daratumumab + Lenalidomide (Active Comparator)
  Interventions: Drug: Daratumumab; Drug: Lenalidomide
- Comparative treatment : Elranatamab + Lenalidomide (Experimental)
  Interventions: Drug: Elranatamab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Elranatamab — Each injection may be up to 2 mL in volume; however, if the maximum volume allowed per institution's policy is lower than 2 mL, the number of injections may be increased to accommodate this difference in volume and ensure the correct dose is delivered. Elranatamab should be administered to the abdomen, with preference given to the lower quadrants when possible.
  Each participant may receive study intervention for a maximum of 24 cycles.
  Arms: Comparative treatment : Elranatamab + Lenalidomide
Drug: Daratumumab — 1800 mg will be administrated every cycles
  Arms: Usual care : Daratumumab + Lenalidomide
Drug: Lenalidomide — Daily administarted during 21 days, at each cycle

SUMMARY:
Lenalidomide is a standard of care for maintenance therapy after autologous stem cell transplantation in newly diagnosed myeloma patients. Recently, two large phase 3 randomized trials demonstrated a progression free survival benefit with daratumumab maintenance post autologous stem cell transplantation. Bispecific antibodies targeting B-Cell Maturation Antigen are approved for the treatment of relapsed refractory myeloma patients after 3 prior lines of therapy including proteasome inhibitor, immunomodulator IMiD and anti CD38 monoclonal antibody. In the cohort A of the MAGNETISMM-3 phase 2 study (n=123), elranatamab single-agent demonstrated strong efficacy with favorable safety profile in patients with advanced multiple myeloma (median of 5 prior lines, 96% of patients with triple class refractory disease). Lenalidomide has been shown to promote cytotoxic activity of CD3 bispecific antibodies. 7We propose a phase 2 randomized study comparing elranatamab plus lenalidomide versus daratumumab plus lenalidomide for 2 years as post-transplant maintenance in patients with newly diagnosed multiple myeloma. The primary objective is minimal residual disease rate after one year of maintenance. Secondary objectives include Progression-Free Survival, safety, quality of life, return to work and overall survival.

DETAILED DESCRIPTION:
Post transplant maintenance with daratumumab and lenalidomide is now considered a standard of care in transplant eligible newly diagnosed myeloma patients. The T-cell engager elranatamab is approved for relapsed myeloma patients, and is currently evaluated in frontline therapy. The combination of bispecific antibody with lenalidomide demosntrated promising response rates with favorable safety profile.

The phase 2 randomized study ELMMA aims to compare the efficacy and safety of elranatamab plus lenalidomide verus daratumumab plus lenalidomide for 2 years as post-transplant maintenance in newly diagnosed myeloma patients.

Target population: n=176, newly diagnosed myeloma transplant eligible following 4-6 cycles of quadruplet induction and autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. - Male or female subjects, 18 years of age or older
2. - Voluntary written informed consent must be given before performance of any study-related procedure not part of normal medical care, with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.
3. - Subject must have documented multiple myeloma according to International Myeloma Working Group (IMWG) criteria and have received 4 to 6 cycles of quadruplet-based therapy including proteasome inhibitor, IMID and anti CD38 monoclonal antibody.
4. - Subject must have received only one line of therapy and achieved at least a partial response as per IMWG 2016 criteria.
5. - Subject must have received high-dose melphalan and ASCT within 12 months of the start of induction therapy and be within 6 months of the last ASCT at the time of first treatment dose.
6. - Subject must have NGS analysis performed at time of MM diagnosis and/or adequate stored bone marrow material allowing NGS analysis (IUCT-Oncopole, Toulouse, France) in order to calibrate MRD analysis.
7. - Karnofsky performance status score ≥ 50% (eastern cooperative oncology group performance status ECOG score ≤ 2).
8. - Subject must have clinical laboratory values meeting the following criteria during the Screening Phase:

   * Hematology : Hemoglobin >8.0 g/dL without prior RBC transfusion within 7 days before the laboratory test; recombinant human erythropoietin use is permitted) + Platelets ≥75×109/L (without transfusion support or thrombopoietin receptor agonist within 7 days before the laboratory test) + Absolute neutrophil count ≥1.0×109/L (prior growth factor support is permitted but must be without support for 7 days for G-CSF or 14 days for pegylated-G-CSF)
   * Chemistry : AST and ALT ≤2.5× upper limit of normal (ULN) + CrCl ≥30 mL/min based on Cockroft-Gault formula calculation or a 24-hour urine collection + Total bilirubin ≤1.5×ULN; except in participants with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin ≤1.5×ULN is required) + Serum calcium corrected for albumin ≤14 mg/dL (≤3.5 mmol/L)
9. - Women of childbearing potential must have a negative serum or urine pregnancy test within 10 to 14 days prior to therapy and repeated within 24 hours before starting study drug. They must commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control (One highly effective method and one additional effective method) used at the same time, beginning at least 4 weeks before initiation of lenalidomide treatment and continuing for at least 6 months after the last dose of Lenalidomide or Elranatamab depending on the last treatment taken. Highly effective contraceptive methods are defined as any of the following methods: combined hormonal contraception (containing estrogen and progestin) combined with ovulation inhibition (oral, intravaginal, transdermal), progestin-only hormonal contraception combined with ovulation inhibition (oral, injectable, implantable), intrauterine device (IUD), hormone-releasing intrauterine system (IUS), bilateral tubal occlusion, vasectomised partner, sexual abstinence.Women must also agree to notify pregnancy during the study.
10. - Men must agree to not father a child and agree to use a latex condom during therapy and for 6 months after the last dose of study drug, even if they have had a successful vasectomy, if their partner is of childbearing potential.

Exclusion Criteria:

1. - Subjects have received any prior anti BCMA therapy.
2. - Subject have received post transplantation maintenance therapy.
3. - Subject intolerant to lenalidomide or have discontinued treatment due to any AE related to lenalidomide.
4. - Subject is exhibiting clinical signs of meningeal involvement of multiple myeloma.
5. - Myocardial infarction within 6 months prior to enrollment according to NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
6. - Uncontrolled hypertension.
7. - Subjects with known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 < 50% of predicted normal.
8. - Subjects with a history of moderate or severe persistent asthma within the past 2 years, or with uncontrolled asthma of any classification at the time of screening (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
9. - Subject has plasma cell leukemia (according to WHO criterion: ≥ 20% of cells in the peripheral blood with an absolute plasma cell count of more than 2 × 109/L) or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
10. - Systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study treatment.
11. - Known intolerance to steroid therapy.
12. - History of allergy to any of the study medications, their analogues, or excipients in the various formulations.
13. - Subject has had major surgery within 2 weeks before randomization or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study. Kyphoplasty or Vertebroplasty are not considered major surgery.
14. - Clinically relevant active infection or serious co-morbid medical conditions.
15. - Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer free of disease since 5 years.
16. - Female subject who is pregnant or breast-feeding.
17. - Serious medical or psychiatric illness likely to interfere with participation in study.
18. - Uncontrolled diabetes mellitus.
19. - Active HBV, HCV, SARS-CoV-2, HIV, or any active, uncontrolled bacterial, fungal, or viral infection. Active infections must be resolved at least 21 days prior to enrollment. Treatment with systemic anti-infective agents must have completed at least 28 days prior to enrollment. Prophylactic use of systemic agents is permitted.

    * COVID-19/SARS-CoV-2: SARS-CoV-2 PCR testing is mandated within 5 days prior to enrollment. Participants with positive PCR test result for SARS-CoV-2 within 5 days prior to enrollment, or suspected of having SARS-CoV-2, are excluded.
    * HIV: In equivocal cases, participants whose viral load is negative may be eligible. HIV seropositive participants who are otherwise healthy and at low risk for AIDS-related outcomes could be considered eligible. Potential eligibility for a specific HIV positive protocol candidate should be evaluated and discussed with the sponsor prior to screening, considering current and past CD4+ and T-cell counts, history (if any) of AIDS defining conditions (eg, opportunistic infections), status of HIV treatment and the potential for drug-drug interactions.
    * HBV:

      * Participants with a positive HBsAg test (ie, either acute or chronic active hepatitis) are excluded.
      * Participants with HBV antibody positivity indicating immunity, either due to vaccination or prior natural infection, are eligible.
      * Participants with positive anti-HBcAb but negative HBsAg and negative anti-HBsAb profile are eligible if HBV DNA is not detected.

    For additional details, refer to CDC website (https://www.cdc.gov/hepatitis/HBV/PDFs/SerologicChartv8.pdf).

    • HCV: Positive HCV antibody is indicative of infection but may not necessarily render a potential candidate ineligible, depending on clinical circumstances. If exposure to HCV is recent, HCV antibody may not have yet turned positive. In these circumstances it is recommended to test for HCV RNA. If HCV RNA is detected, the patient is not eligible. Refer to CDC website for further details(https://www.cdc.gov/hepatitis/hcv/pdfs/hcv_graph.pdf).
20. - Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs.
21. - Subjects unable or unwilling to undergo antithrombotic prophylactic treatment.
22. - Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease negativity rate | At the beginning of cycle 13 (each cycle is 28 days)
  Minimal Residual Disease negativity rate (10-6, NGS) status after 12 cycles of maintenance

SECONDARY OUTCOMES:
Safety and tolerability of Dara-Len and Elra-Len | 4 years
  Presence and severity of Treatment-Emergent Adverse Events defined by National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (Number of Treatment-Emergent Adverse Events), except for Cytokine Release Syndrome and Immune effector Cell-Associated Neurotoxicity syndrome, which will be assessed based on American Society for Transplantation and Cellular Therapy guidelines.
Progression-free survival | 4 years
  Progression-free survival, defined as the time from randomization to the first occurrence of Progressive Disease, or death from any cause, whichever occurs first. Subjects alive and for whom disease progression has not been observed will be censored at the last date of follow-up.
Minimal Residual Disease negativity with the threshold evaluated at one year after randomisation | At the beginning of cycle 13 (each cycle is 28 days)
  Rate of Minimal Residual Disease status at one year after randomisation
Minimal Residual Disease negativity with the threshold evaluated at one two years | At the beginning of cycle 25 (each cycle is 28 days)
  Rate of Minimal Residual Disease status at two years after randomization
Sustained Minimal Residual Disease negativity | At the beginning of cycle 13 and 25 (each cycle is 28 days)
  Rate of patients with Minimal Residual Disease negative status during at least 12 months (at least two consecutive times)
Complete Response or better | 4 years
  The rate of complete response or better as defined by International Myeloma Working Group 2016
Overall survival | 4 years
  Time from randomisation to the date of death due to any cause. Subjects alive will be censored at the last date of follow-up.
Progression-free survival 2 | 4 years
  Time from randomization to either second line Progressive Disease (assessed by investigator on the first subsequent line of antimyeloma therapy) or death, whichever occurs first. Subjects alive and for whom a second disease progression has not been observed will be censored at the last date of follow-up.
Ability of return to work | At the beginning of cycle 1 (each cycle is 28 days), at 3 months, 6 months, 12 months, 24 months, 36 months and 48 months
  Ability of return to work assessed by a specific questionnaire

OTHER OUTCOMES:
Determine biological prognostic factors influencing Minimal Residual Disease | At screnning (Baseline)
  Value of biological prognostic factors (ISS Stage, Cytogenetics)
Determine biological prognostic factors influencing complete response. | At screnning (Baseline)
  Value of biological prognostic factors (ISS Stage, Cytogenetics)
Descriptive quality of life | At Screening, At the beginning of every 3 cycles (each cycle is 28 days), at the beginning of cycle 24, and during the Follow-Up before Progressive Disease
  Descriptive quality of life assessed by EQ-5D-5L and EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (36):
- France (36):
  - CHU Angers, Angers
  - CH Côte Basque, Bayonne
  - CHU Besançon, Besançon
  - CHU Caen, Caen
  - Hôpital d'Instruction des Armées Percy, Clamart
  - CHU Clermont- Ferrand - Hôpital ESTAING, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - CHRU Dijon, Dijon
  - Institut de cancérologie de Bourgogne, Dijon
  - Hôpital Annecy Genevois, Épagny
  - CHD Vendée, La Roche-sur-Yon
  - CH Le Mans - Centre de cancérologie de la Sarthe, Le Mans
  - CH de Libourne, Libourne
  - CHU Limoges, Limoges
  - Groupement Hospitalier Bretagne Sud, Lorient
  - Centre Léon BERARD, Lyon
  - IPC Marseille, Marseille
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU de Nice - Hôpital l'Archet 1, Nice
  - CHU de Nîmes - Institut de Cancérologie du Gard, Nîmes
  - Hopital St Louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Hôpital St Antoine, Paris
  - CH Saint-Jean, Perpignan
  - CHRU - Hôpital du Haut Lévêque, Pessac
  - CH Périgueux, Périgueux
  - CHU de Poitiers, Poitiers
  - CH Cornouaille Quimper, Quimper
  - CH de Saint Nazaire, Saint-Nazaire
  - ICANS, Strasbourg
  - CH Tarbes-Lourdes, Tarbes
  - CHU Toulouse, Toulouse
  - CHRU Bretonneau, Tours
  - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: Undecided